CLINICAL TRIAL: NCT04609488
Title: An Exploratory Study to Assess Surfactant Levels in COVID-19 Patients Who Will be on Ventilatory Support Due to Severe Respiratory Failure
Brief Title: Surfactant Levels in the Lungs of COVID-19 Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Henning Bay Nielsen, MD DMSci adj Professor specialist consultant Anesthesia, Zealand University Hospital
Other Study IDs: SJ-859x
Record Dates: First submitted 2020-10-28; First posted 2020-10-30 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: To Assess Surfactant Levels in Lung Fluid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tracheal fluid
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID
  Interventions: Diagnostic Test: Surfactant assessment
- non-COVID
  Interventions: Diagnostic Test: Surfactant assessment

INTERVENTIONS:
Diagnostic Test: Surfactant assessment — To determine surfactant levels in lung fluid

SUMMARY:
NAME of STUDY: Surfactant levels in the lungs of COVID-19 patients BACKGROUND

* Infection with SARS-CoV-2 may induce respiratory failure.
* COVID-19 associated respiratory failure may require ventilatory support.
* SARS-CoV-2 uses alveolar type II cells for virus replication.
* Alveolar type II cells are responsible for surfactant production and lack of surfactant causes respiratory failure in preterm neonates.
* Lack of surfactant may play role for respiratory failure in COVID-19 patients DESIGN Exploratory prospective study design without therapeutic intervention of any kind. Lung fluid will be donated as part of standard care procedures.

HYPOTHESIS Surfactant is measurable in tracheal secretions by mid-infrared FTIR spectroscopy determined surfactant spectra. Surfactant is reduced in COVID-19 patients requiring ventilator support as compared to non- COVID-19 patients. Dysfunctional surfactant in COVID-19 patients regain its function when respiratory function improves.

POPULATION Main population is patients with COVID-19 pneumonia that requires ventilatory support.

OUTCOME MEASURES Primary outcome is the level of surfactant in lung fluid as obtained by tracheal suction.

SAMPLE SIZE In total 30 patients will be included: twenty COVID-19 patients and 10 non-COVID-19 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients positive for coronavirus 2 (SARS-CoV-2) AND
2. Respiratory failure requiring mechanical ventilation support OR respiratory failure requiring oxygen supplementation AND
3. Age > 18 years AND
4. Permission from next of kin

Exclusion Criteria:

Inability to obtain TS or BL as determined by clinical judgement by responsible clinician. Patients with known surfactant dysfunction (such as mutations in the SFTPB or ABCA3 gene). Imminent expected death within 24 hours. Stage 4 severe chronic kidney disease or requiring dialysis. Liver failure. Anticipated transfer to another hospital within 72 hours. Participation in another study which in the opinion of the investigator would prevent enrollment for safety purposes.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients are COVID-19 patients requiring ventilatory support by mechanical ventilation as well as Non-COVID-19 patients requiring ventilatory support by mechanical ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Surfactant | Two years
  The primary outcome is surfactant levels in lung fluid

IPD SHARING:
Plan to Share IPD: Undecided